CLINICAL TRIAL: NCT06276855
Title: Associate Professor Registered Nurse Doctor of Philosophy
Brief Title: Sleep Hygiene Education in Individuals With Fibromyalgia; Sleep Quality, Pain and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Tülay Kars Fertelli, Assoc. Prof, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CUtülay
Record Dates: First submitted 2024-01-22; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Fibromyalgia
Keywords: Sleep Hygiene; Sleep Quality; Pain; Depression; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Sleep Hygiene; Sleep Initiation and Maintenance Disorders; Pain; Depression

STUDY DESIGN:
Intervention Model Description: Experimental group Control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The DIF, PSQI, VAS, and BDI were also administered to individuals in the control group during the first interview, but no education was provided to them. The participants were given an appointment to meet at the hospital one month later. At the final polyclinic appointment one month later, the VAS, PSQI, and BDI were administered for the second time and took an average of 15-20 minutes to complete. In line with ethical principles, they were provided with individual education on sleep hygiene and sleep hygiene education booklets at the final polyclinic appointment. The same researcher collected the data and provided the education to avoid bias.
- Experimental group (Experimental): During the first interview, the DIF, PSQI, VAS, and BDI were administered to individuals in the experimental group. Each education session lasted an average of 30 minutes and was conducted face-to-face. Sleep hygiene education booklets were provided to individuals at the end of the education session. Studies suggest that at least one month should pass for behavioral change to occur after the education session. Therefore, the participants were given an appointment to meet at the hospital one month later. At the final interview one month after the education, the VAS, PSQI, and BDI were administered for the second and final time and took an average of 15-20 minutes to complete.
  Interventions: Other: Sleep hygiene education

INTERVENTIONS:
Other: Sleep hygiene education — The sleep hygiene education booklet was prepared by the researchers by in line with the literature. The booklet contains information on the definition and benefits of sleep, sleep problems during insomnia, arrangements for regular sleep, and the principles of sleep hygiene. The principles of sleep hygiene include individual habits that facilitate sleep, proper arrangement of the physical environment, exercises before going to bed, and dietary habits. This educational content was applied to those in the experimental group. The education took an average of 30 minutes.
  Arms: Experimental group

SUMMARY:
Objective: This semi-experimental study was conducted to determine the effect of sleep hygiene education on sleep quality, pain, and depression in individuals with fibromyalgia.

Patients and methods: A sample of 70 individuals with fibromyalgia (35 experimental, 35 control) were included in the study. Data was collected using the Pittsburgh Sleep Quality Index, the Visual Analog Scale, and the Beck Depression Inventory.

DETAILED DESCRIPTION:
Objective: This semi-experimental study was conducted to determine the effect of sleep hygiene education on sleep quality, pain, and depression in individuals with fibromyalgia.

Background: Sleep problems, pain, and depression are common health issues in individuals with fibromyalgia. However, studies on sleep hygiene education to address these problems are limited in the literature.

Methods: A sample of 70 individuals with fibromyalgia (35 experimental, 35 control) were included in the study. Data was collected using the Pittsburgh Sleep Quality Index, the Visual Analog Scale, and the Beck Depression Inventory.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for the study were as follows:

* Being 18 years of age or older,
* Having a diagnosis of Fibromyalgia (FM) for at least 3 months,
* Being reachable,
* Agreeing to participate in the study,
* Not receiving treatment for depression,
* Not having received similar education on sleep hygiene,
* Having a VAS pain score >3,
* Having a PSQI score >5.

Exclusion Criteria:

Additionally, the exclusion criteria for the study were as follows:

* Having a diagnosis of FM for less than 3 months,
* Using sleep medication,
* Having chronic illnesses that could interfere with sleep such as Chronic Obstructive Pulmonary Disease (COPD) or asthma,
* Working on night shifts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Demographic Information Form (DIF). | 1 month
  This form was prepared by the researcher based on the literature and consists of 10 questions about the FM patients' sociodemographic and disease characteristics (age, gender, educational status, etc.).
Pittsburgh Sleep Quality Index (PSQI). | 1 month
  The PSQI evaluates the quality of sleep in the last month. It consists of 19 items and 7 components. Each item is evaluated on a 0-3 point scale, and the sum of scores from seven components gives the total PSQI score. The total score ranges from 0 to 21. A high total score indicates poor sleep quality. A total PSQI score of ≤5 indicates "good sleep," while a score of >5 indicates "poor sleep." The Cronbach's alpha value of the scale is 0.80. In this study, the Cronbach's alpha was found to be 0.83.
Visual Analog Scale (VAS). | 1 month
  The VAS is a valid and reliable scale to measure the intensity of chronic pain. It is rated from "0 = no pain" to "10 = worst possible pain". The intervals for pain intensity are <3 for mild pain, 3-6 for moderate pain, and >6 for severe pain. The Cronbach's alpha value of the scale is 0.97. In this study, the Cronbach's alpha was found to be 0.92.
Beck Depression Inventory (BDI). | 1 month
  The scale consists of a total of 21 items. The highest possible total score is 63. A high total score indicates a higher level of depression. The severity of depression is categorized as follows: 0-9 = minimal, 10-16 = mild, 17-29 = moderate, and 30-63 = severe depression. The internal consistency coefficient of the scale is 0.86. In this study, the Cronbach's alpha was found to be 0.83.

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet University, Sivas, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No